CLINICAL TRIAL: NCT02321059
Title: Validation of the Goodstrength System for Assessment of Abdominal Wall Strength in Patients With Incisional Hernia
Acronym: VAGSI
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kristian Kiim Jensen, MD, Bispebjerg Hospital
Other Study IDs: H-1-2014-008
Record Dates: First submitted 2014-11-11; First posted 2014-12-22 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Incisional Hernia
Keywords: incisional hernia; hernia; abdominal wall strength; validation; physical activity
MeSH Terms: conditions — Incisional Hernia; Hernia; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No incisional hernia group: Healthy volunteers with an intact abdominal wall.
  Interventions: Device: Measurement of abdominal wall strength
- Incisional hernia group: Patients with a ventral incisional hernia.
  Interventions: Device: Measurement of abdominal wall strength

INTERVENTIONS:
Device: Measurement of abdominal wall strength — Test-retest examination of the reliability of the Goodstrength trunk dynamometer

SUMMARY:
Patients with an incisional hernia in the midline and controls with an intact abdominal wall are examined twice with one week apart, in order to establish the test-retest reliability and internal and external validity of the Goodstrength trunk dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score 1-3
* Age equal to or above 18
* Ventral incisional hernia OR intact abdominal wall

Exclusion Criteria:

* Pregnancy
* Severe heart disease (New York Heart Association class III-IV)
* Severe pulmonary disease
* Severe musculoskeletal disease
* Systemic treatment with glucocorticoid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients on waiting list for repair of a ventral incisional hernia and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Abdominal wall strength measured by the Goodstrength system | One week
  Change in abdominal wall strength from baseline to follow-up.

SECONDARY OUTCOMES:
Physical activity the last week, assessed by the International Physical Activity Questionnaire | Once, at baseline examination
Self-assessed abdominal wall strength, as measured on a visual analogue scale | Once, at baseline examination
Trunk extensor strength measured by the Goodstrength system | One week
  Change in trunk extensor strength from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian K Jensen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Copenhagen, Denmark